CLINICAL TRIAL: NCT04762719
Title: Dynamic Positron Emission Tomography Imaging With 11C-ER176 to Delineate Macrophage Activation in Diabetic Gastroparesis
Brief Title: PET Imaging to Delineate Macrophage Activation in Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Madhusudan (Madhu) Grover, MBBS, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-010260
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Gastroparesis With Diabetes Mellitus
Keywords: macrophages, immune cells, gastric emptying, gastroparesis, imaging
MeSH Terms: conditions — Diabetes Mellitus; Gastroparesis

STUDY DESIGN:
Intervention Model Description: Three groups of patients (diabetic; diabetic gastroparesis; healthy volunteers) will undergo PET-CT. The diabetic gastroparesis group will also undergo gastric muscle biopsy of the involved and uninvolved area to validate immune changes visualized on imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Diabetic Gastroparesis Subjects (Experimental): Type I or II diabetes subjects who also have a diagnosis of Gastroparesis (defined by gastric retention of Tc-99m >20% at 4 hrs on scintigraphy). Subjects will receive PET/CT Scan with 11C-ER176 and a core biopsy of gastric muscle
  Interventions: Drug: PET/CT Scan with 11C-ER176; Diagnostic Test: Core biopsy of gastric muscle
- Diabetic without gastroparesis subjects (Experimental): Type I or II diabetes subjects who have not been clinically diagnosed with Gastroparesis. Subjects will receive PET/CT Scan with 11C-ER176
  Interventions: Drug: PET/CT Scan with 11C-ER176
- Healthy Subjects (Placebo Comparator): Healthy subjects will be age-matched and receive a PET/CT Scan with 11C-ER176
  Interventions: Drug: PET/CT Scan with 11C-ER176

INTERVENTIONS:
Drug: PET/CT Scan with 11C-ER176 — Subjects will have a low-dose, non-gated, non-contrast-enhanced, free-breathing CT from the orbits to upper thigh for attenuation correction (CTAC) and anatomic co-localization. Immediately following the start of the PET scan, 518 MBq (14 mCi) (range 370-666 MBq; 10-18 mCi) of 11C-ER 176 will be administered intravenously followed by a saline flush. A whole-body PET scan from the orbits to upper thigh will then be acquired.
Diagnostic Test: Core biopsy of gastric muscle — The echoendoscope (Aloka Arietta 850; Olympus, Center Valley, PA) will be advanced into the gastric lumen and a site targeted for EUS-guided core biopsies based on findings of the PET scan. Fine needle biopsy of the gastric wall will be performed.
  Arms: Diabetic Gastroparesis Subjects

SUMMARY:
Macrophage-driven immune dysregulation has been shown to be involved in pathophysiology of diabetic gastroparesis. Currently, there are no non-invasive ways to study macrophage activation in humans. The researchers are trying to determine the utility of 11C-ER176 based PET-CT scanning to determine pro-inflammatory macrophage activation in gastric wall of patients with diabetic gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 70 years of age.
* Ability to provide informed consent.
* Type I or II diabetes mellitus.
* Gastroparesis defined by gastric retention of Tc-99m > 60 % at 2 hrs and/or > 10% at 4 hours on scintigraphy.
* Average Gastroparesis Cardinal Symptom Index (GCSI) ≥ 3 indicating moderate-severe symptoms.

Exclusion Criteria:

* Women who are pregnant or cannot stop breast feeding for 24 hours.
* Using anti-coagulants, anti-inflammatory medications (NSAIDs, corticosteroids, etc.) or immunosuppressive therapies within the 4 weeks prior.
* Opioid use within the last 4 weeks of gastric emptying scintigraphy.
* Prior gastric surgery.
* History of IBD, celiac disease, eosinophilic gastroenteritis, microscopic colitis.

Healthy Subjects Exclusion criteria

* no clinical history of diabetes or any GI symptoms
* no inflammatory disorders of the GI tract
* no use of anti-inflammatory or immunosuppressive therapies

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Gastroparesis Subjects: Type I or II diabetes subjects who also have a diagnosis of Gastroparesis (defined by gastric retention of Tc-99m >20% at 4 hrs. on scintigraphy), received a PET/CT scan with 11C-ER176 and a core biopsy of gastric muscle.
  PET/CT scan with 11C-ER176: Subjects received a low-dose, non-gated, non-contrast-enhanced, free-breathing CT from the orbits to upper thigh. Immediately following the start of the PET scan, 518 MBq (14 mCi) (range 370-666 MBq; 10-18 mCi) of 11C-ER 176 was administered intravenously followed by a saline flush. A whole-body PET scan from the orbits to upper thigh was then acquired.
  Core biopsy of gastric muscle: The echoendoscope (Aloka Arietta 850; Olympus, Center Valley, PA) was advanced into the gastric lumen and a site targeted for EUS-guided core biopsies based on findings of the PET scan. Fine needle biopsy of the gastric wall was performed.
- Diabetic Without Gastroparesis Subjects: Type I or II diabetes subjects who have not been clinically diagnosed with Gastroparesis. Subjects received a PET/CT scan with 11C-ER176.
  PET/CT scan with 11C-ER176: Subjects received a low-dose, non-gated, non-contrast-enhanced, free-breathing CT from the orbits to upper thigh. Immediately following the start of the PET scan, 518 MBq (14 mCi) (range 370-666 MBq; 10-18 mCi) of 11C-ER 176 was administered intravenously followed by a saline flush. A whole-body PET scan from the orbits to upper thigh was then acquired.
- Healthy Subjects: Healthy subjects were age-matched and received a PET/CT scan with 11C-ER176.
  PET/CT scan with 11C-ER176: Subjects received a low-dose, non-gated, non-contrast-enhanced, free-breathing CT from the orbits to upper thigh. Immediately following the start of the PET scan, 518 MBq (14 mCi) (range 370-666 MBq; 10-18 mCi) of 11C-ER 176 was administered intravenously followed by a saline flush. A whole-body PET scan from the orbits to upper thigh was then acquired.
Period: Overall Study
Arm/Group | Diabetic Gastroparesis Subjects | Diabetic Without Gastroparesis Subjects | Healthy Subjects
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetic Gastroparesis Subjects | Diabetic Without Gastroparesis Subjects | Healthy Subjects | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (7.0) | 48.0 (13.0) | 47.0 (11.0) | 48.0 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 3 | 4 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Uptake of 11C-ER 176 in the Stomach Muscle
Description: All patients will have a PET/CT with 11C-ER 176. On each PET image, volumes of interest areas will be drawn around the stomach and other organs that may show radiotracer accumulation. The uptake of radiotracer 11C-ER 176 in each area will be quantified and reported as maximum standardized uptake values (SUVmax)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Diabetic Gastroparesis Subjects | Diabetic Without Gastroparesis Subjects | Healthy Subjects
Number analyzed (Participants) | 4 | 4 | 4
SUVmax
  stomach pylorus | 5.5 (1.0) | 8.4 (4.1) | 4.6 (0.2)
  stomach gastric fundus | 7.8 (1.9) | 13.1 (8.3) | 9.0 (1.6)
  stomach body | 7.8 (1.9) | 13.0 (9.2) | 7.7 (1.9)
  duodenum | 7.0 (1.8) | 9.5 (6.8) | 6.2 (2.1)

2. Secondary Outcome: Percentage of Immune Cells With CD45 Expression
Description: An upper endoscopy procedure was done for diabetic gastroparesis patients and full thickness core tissue samples were taken in the stomach in areas that demonstrated 11C-ER 176 uptake in the PET scan as well as non-enhancing control areas. Cytometry by time of flight (CyTOF) mass spectrometry system was used to determine the proportions of immune cell types with CD45.
Time Frame: baseline
Population: The tissue obtained from diabetic gastroparesis group was not of sufficient size or volume to perform quantitative (%) assessment. Outcome measure for diabetic gastroparesis subjects only.
Arm/Group | Diabetic Gastroparesis Subjects | Diabetic Without Gastroparesis Subjects | Healthy Subjects
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from baseline to end of study, approximately 14 days.
Arm/Group | Diabetic Gastroparesis Subjects | Diabetic Without Gastroparesis Subjects | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 0/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetic Gastroparesis Subjects (N=4) | Diabetic Without Gastroparesis Subjects (N=4) | Healthy Subjects (N=4)
Sore throat (Gastrointestinal disorders) | 1 | 0 | 0
Uvular abrasion (Gastrointestinal disorders) | 1 | 0 | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/19/NCT04762719/Prot_SAP_001.pdf